CLINICAL TRIAL: NCT01914354
Title: Role of CD28null NKG2Dpos T Cells on Human Alloimmune Reactivity: An Untargeted T Cell Population" (# 859869783).
Brief Title: Role of CD28null NKG2Dpos T Cells on Human Alloimmune Reactivity T Cell Population
Acronym: NKG2D
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 859869783
Record Dates: First submitted 2012-01-19; First posted 2013-08-02 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Kidney Transplant
Keywords: T cells; Human Alloimmune Reactivity; immunosuppression

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples Without DNA — blood/serum
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational multi-center study to determine whether any single immune monitoring test or a combination of tests obtained in the first 6 months after renal transplantation correlates with acute rejection or graft loss in renal allograft recipients receiving commonly used immunosuppressive.

ELIGIBILITY:
Inclusion Criteria:

* human kidney transplant recipients
* ATG or basiliximab induction therapy

Exclusion Criteria:

* induction therapy other than ATG or basiliximab

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cohort of 80 living and deceased donor kidney transplant recipients and 10 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To document the prevalence and frequencies of CD4+ and CD8+ CD28null/NKG2Dpos T cells at the time of transplantation. | 6 months
To test whether CD28null/NKG2Dpos T cells have unique rapid activation properties to allogeneic HLA antigens in vitro | 6 months

SECONDARY OUTCOMES:
To study the clinical correlations between the frequencies of alloreactive CD28null/NKG2Dpos T cells with kidney graft function and histopathology. | 6 months
To test the effects of induction therapy with rabbit anti-thymocyte globulin (ATG) vs. IL-2 receptor blocker antibodies on circulating CD28null/NKG2Dpos T cells. | 6 months